CLINICAL TRIAL: NCT07093255
Title: A Phase 1b, Dose Escalation Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of FLQ-101 in Premature Neonates at High Risk of Developing ROP
Brief Title: Safety, PK and PD of FLQ-101 in Premature Neonates
Acronym: tROPhy-1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: FELIQS INC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLQCT-01
Record Dates: First submitted 2025-07-16; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Retinopathy of Prematurity (ROP)
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FLQ-101 (Experimental)
  Interventions: Drug: FLQ-101

INTERVENTIONS:
Drug: FLQ-101 — The invervention comprises 3 Groups:
  * Group 1: Low Dose
  * Group 2: Middle Dose
  * Group 3: High Dose

SUMMARY:
The purpose of this study is to evaluate safety and efficacy outcomes following exposure to FLQ-101.

ELIGIBILITY:
Inclusion Criteria:

* Written consent is obtained from parent(s) or legal guardian.
* Neonates born at 26 weeks +0 days and 27 weeks +6 days of gestation.
* Male or female infants with a birth weight greater than or equal to 650 gm.

Exclusion Criteria:

* Neonates with congenital malformation of the eye or any other ocular condition that may prevent or relevantly affect any of the assessments or procedures.
* Neonates with serious congenital anomalies, severe congenital infection, and chromosomal abnormalities.
* Neonates who are seriously ill and not expected to survive.
* Neonates with heart disease, including cardiomyopathy, serious arrhythmias, and congenital heart disease. (Neonates with patent foramen ovale may be included in the study if clinically stable).
* Neonates that are small for gestational age defined as having a weight <10th percentile at birth based on the Fenton growth charts for gestational age and sex.
* Neonates with history of or ongoing intraventricular hemorrhage (IVH) grades 2, 3 or 4. Neonates with IVH grade 1 may be included in the study at the discretion of the PI.
* Neonates with any other medical conditions or clinically significant comorbidities or circumstances that in the opinion of the investigator may have a relevant impact on study participation or any of the study assessments or procedures.
* Infants scheduled to participate in other interventional clinical trials while participating in the study and until reaching end of study.

Ages: 4 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events | Day 1 to 36 weeks PMA(post menstrual age)

SECONDARY OUTCOMES:
Pharmacokinetic parameters of FLQ-101 | Day 1 to 24 hours post first oral dose
Pharmacodynamic parameters of FLQ-101 | Day 1 to 24 hours post first oral dose

IPD SHARING:
Plan to Share IPD: Undecided